CLINICAL TRIAL: NCT02576106
Title: Evaluation of Percutaneous Treatment by Cryoablation of Unifocal Invasive Breast Carcinoma in Menopausal Women With Indication of Lumpectomy
Acronym: CRYOSE01
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Leon Berard (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ET15-001
Record Dates: First submitted 2015-10-12; First posted 2015-10-15 (Estimated); Last update posted 2020-10-22 (Actual); Status verified 2018-08

CONDITIONS: Carcinoma, Ductal, Breast; Menopausal
MeSH Terms: conditions — Carcinoma, Ductal, Breast | interventions — Cryosurgery; Cryotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Cryoablation (Experimental): Cryoablation of the tumor followed by a lumpectomy as practiced in standard care
  Interventions: Device: Cryoablation

INTERVENTIONS:
Device: Cryoablation
  Other Names: Cryotherapy

SUMMARY:
The primary objective of this monocentric and feasibility study is to review the efficacy of cryotherapy in the treatment of unifocal mammary carcinomas in post-menopausal patients, with lumpectomy indication.

The efficacy is defined by the rate of success of cryotherapy procedures. For each one of those evaluated process, an success will be defined on the tumor sample of lumpectomy by the absence of viable tumour cells.

On the basis of our expertise, it seems interesting to propose this experimental procedure to patients as described above.

ELIGIBILITY:
Inclusion Criteria:

* Non inflammatory unilateral and unifocal breast cancer with indication of lumpectomy
* Menopausal women with age > 55 years
* Tumor size <= 15 mm by ultrasonography
* Histological confirmation (by biopsy) of invasive ductal carcinoma with SBR (Scarff-Bloom-Richardson) grade (modified by Ellis & Elston) 1 or 2; hormone receptors positive (Estrogen Receptor and/or Progesterone Receptor) and negative Human epidermal growth factor receptor (HER2)
* Good lesion boundary with ultrasonography and MRI
* Minimal distance of 5 mm between the skin and the tumor
* Performance Status 0-1
* Ability to understand and willingness to sign a written informed consent document
* Covered by a medical insurance
* Signed informed consent

Exclusion Criteria:

* Invasive lobular carcinoma
* Tumor with retro-nipple location
* Extended microcalcifications (> 15 mm) with mammography
* Xylocaine allergy
* Patient deprived of freedom

Min Age: 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2020-01 (Actual); Study Completion 2020-01 (Actual)

PRIMARY OUTCOMES:
The rate of success of cryoablation procedure | 45 days after cryoablation
  percentage of viable cells in the piece of lumpectomy

CONTACTS AND LOCATIONS:
Overall Officials: Frank Pilleul, MD-PhD, Principal Investigator — Centre Leon Berard
Locations (1):
- Centre Léon Bérard, Lyon, France